CLINICAL TRIAL: NCT07339605
Title: Clinical and Radiographic Outcomes After Flapless Approach of Intrabony Defects With the Application of Enamel Matrix Derivative Versus Hyaluronic Acid: A Randomized Controlled Clinical Trial
Brief Title: Flapless Periodontal Regeneration Using Hyaluronic Acid Versus Enamel Matrix Derivative
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Andres Lopez Roldan, Assistant Professor with PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-ODON-3018356
Record Dates: First submitted 2025-06-30; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-06

CONDITIONS: Guided Tissue Regeneration, Periodontal / Methods; Dental Enamel Proteins* / Therapeutic Use; Alveolar Bone Loss* / Therapy; Hyaluronic Acid* / Therapeutic Use; Humans; Intrabony Defect; Flapless
Keywords: Periodontitis; Intrabony defect; Hyaluronic acid; Enamel matrix derivative; Periodontal regeneration
MeSH Terms: conditions — Alveolar Bone Loss; Periodontitis | interventions — Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- (MINST + NaOCl) + HA (Experimental)
  Interventions: Procedure: Flapless instrumentation of the defect following MINST in conjuction with NaOCl and hyaluronic acid application
- (MINST + EDTA) + EMD (Active Comparator)
  Interventions: Procedure: Flapless instrumentation of the defect following MINST, root conditioning with EDTA and EMD application
- MINST (Sham Comparator)
  Interventions: Procedure: Flapless instrumentation of the defect and product application simulation

INTERVENTIONS:
Procedure: Flapless instrumentation of the defect following MINST in conjuction with NaOCl and hyaluronic acid application — The NaOCL gel buffered with amino acids will be carefully injected and maintained for 60 seconds. Following this, pocket debridement will be carried out following the MINST technique. In order to allow for optimal root visualization and gain access to the intrabony defect, a microsurgical dental mirror will be used in conjunction with an atraumatic gingival retractor for a gentle lateral papilla displacement. Teeth will be instrumented until no residual calculus could be detected after a careful root evaluation with a periodontal explorer and no debris or biofilm flushed out of the pocket after irrigation. If this does not occur, the application of NaOCL, instrumentation and saline solution rinse shall be repeated until this is achieved. After irrigation, sterile gauze will be placed in the vestibule in the proximity of a selected site and a thorough drying of the site will be perfomed with air-spray. HA will be applied with a blunt tipped sterile syringe, until overflowing.
  Arms: (MINST + NaOCl) + HA
Procedure: Flapless instrumentation of the defect following MINST, root conditioning with EDTA and EMD application — Subgingival instrumentation will be performed following the MINST technique in conjunction with a microsurgical dental mirror and an atraumatic gingival retractor without applying any product previously. Teeth will be instrumented until no residual calculus could be detected and no debris or biofilm flushed out of the pocket after irrigation with sterile saline solution. Following this, it will be dried and the root will be conditioned applying EDTA with a thin blunt tip for 2 minutes to remove the dentin mud layer from the root surfaces. Subsequently, the defect area will be carefully rinsed with water-spray and by 5-s passage of ultrasonic instrument's fine tip in the site with no contact to the root surface. A sterile gauze will be placed in the vestibule in the proximity of a selected site and a thorough drying of the site will be performed with an air-spray. Once bleeding control is achieved, EMD will be applied with a blunt tipped sterile syringe (25G), until overflowing.
  Arms: (MINST + EDTA) + EMD
Procedure: Flapless instrumentation of the defect and product application simulation — Subgingival instrumentation will be performed following MINST and EDT+EMD or NaOCl+HA application will be simulated by inserting the manufacturer's syringes within the pocket, but the defects won't receive any adjunct.
  Arms: MINST

SUMMARY:
The goal of this clinical trial is to radiographically assess the effectiveness of minimally invasive non-surgical technique (MINST) combined with local administration of sodium hypochlorite gel (Perisolv®) and 1.6% cross-linked hyaluronic acid (HA, Hyadent BG®) compared to a neutral formulation of EDTA (Prefgel®) and enamel matrix derivative (EMD, Emdogain® FL) in periodontal regeneration. The main questions it aims to answer are:

* ¿Does the combination of MINST with the local administration of sodium hypochlorite gel and 1.6% cross-linked hyaluronic acid show a potential for periodontal regeneration similar to evaluating clinical and radiographic variables compared to a neutral formulation of EDTA and enamel matrix derivative?
* ¿What is the patient perception and satisfaction with the received treatment?

Researchers will compare A (MINST with Perisolv® + Hyadent BG®), B (MINST with PrefGel® + Emdogain® FL) and C(MINST without any bioactive product).

The sample will be distributed according to the following treatments:

* Experimental group: Scaling and root planing (SRP), MINST with Perisolv® + Hyadent BG®.
* Active comparator group: SRP, MINST with PrefGel® + Emdogain® FL.
* Control group: SRP, MINST without any bioactive product.

Patients will be screened by a first visit in which they will be assigned their periodontal status. If they meet the eligibility criteria, they will be treated according to the EFP clinical guideline for periodontitis treatment: step I and step II.If the periodontal defect persists at the 12-week re-evaluation, patients will be randomised to treatment A, B or C.

After the intervention, all participants will be checked weekly for the first 6 weeks to remove accumulated plaque, and every 3 months for 1 year. Periodontal parameters will be re-evaluated 6 and 12 months after periodontal regenerative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Periodontitis stage III or IV, grade A or B (Tonetti et al., 2017): attachment loss ≥ 5mm, radiographic bone loss extending to to the middle third and beyond, tooth loss ≥4 due to periodontitis, probing depth (PD) ≥ 6mm.
* Older adults ≥ 18 years. The number per sex shall be balanced.
* Plaque index (PI) < 1 following initial periodontal therapy and hygiene instructions.
* Bleeding on probing (BoP) ≤ 10%.
* Only patients with optimal compliance, assessed during etiological therapy, will be selected.
* At least a 2-3 wall interproximal bone defect with a radiographically moderate or deep intrabony defect (≥3mm), PD≥ 6mm using a Williams probe on uniradicular teeth or mandibular molars without furcation involvement after non-surgical periodontal treatment.
* Vital teeth or teeth with well-performed root canal treatment.
* Absence of caries, prosthetic restoration or periapical infection in the tooth to be regenerated.
* Absence of systemic pathology.
* Negative history of pregnancy.
* Signed informed consent.
* The participant is willing and able to comply with the necessary visits for the treatments and evaluations scheduled during the clinical study.

Exclusion Criteria:

* The participant is pregnant, breastfeeding or plans to become pregnant in the next 6 months.
* Smoking ≥10 cigarettes/day.
* Daily alcohol intake > 4U.
* Chronic illness or reduced mental capacity that may influence compliance with the protocol.
* Medications or drugs that alter the patient's healing or with concomitant oral manifestations that, in the opinion of the investigator, could interfere with the assessment of safety or efficacy.
* Systemic diseases that may influence treatment such as diabetes mellitus or rheumatoid disease.
* Allergies to drug compounds.
* Antibiotic intake 3 months prior to the start of the study or systemic condition requiring antibiotic coverage at the time of periodontal treatment.
* Periodontal treatment 6 months prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-26 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone fill | Baseline, 6 and 12 months.
  Depth of the intraosseous defect (B - D); and following the healing period (X - C).
  Bone fill (BF) will be calculated by subtracting the (X - C) measurement recorded at the 6-month and 12-month postoperative review from the depth recorded before the regenerative intervention (B - D).

SECONDARY OUTCOMES:
Clinical attachment level (CAL) gain | Baseline, 6 and 12 months.
  CAL is defined as the distance in millimeters between CEJ and the end of the periodontal pocket. The calculation of the CAL before the intervention and after the intervention will be carried out.
Gingival recession | Baseline, 6 and 12 months.
  Distance (mm) between the CEJ and the gingival margin.
Probing pocket depth (PD) | Baseline,6 and 12 months.
  The probing depth will be measured in six areas (disto-buccal, mediate-vestibular, mesio-buccal, disto-palatal, mid-palatal, and mesio-palatal) of each tooth with a Williams PQ-OW 208 396 probe. It will be use with a pressure of 20 grams that is equivalent to the pressure of dropping the weight of the probe without exerting additional pressu
Bleeding on probing | Baseline, 6 and 12 months.
  The "Full mouth bleeding score" (FMBS) will be calculated based on scores of 0 (no bleeding) or 1 (bleeding) after probing depths are checked. The usual thing is to measure 4 points for each tooth, but the investigators have modified the index and value 6 points per tooth (disto-buccal, mid-buccal, mesio-buccal, disto-palatal, mid-palatal and mesio-palatal).
  The investigators consider that the score is 1 when there is a red dot in the bleeding diagram of the periodontogram and 0 when there is a blank box.
Plaque index | Baseline, 6 and 12 months.
  The plaque will be quantified as follows:
  Score 0 = no plaque Score 1 = A film of plaque adhered to the free gingival margin and the adjacent area of the tooth. The plaque can be seen in situ only after the application of a plaque revealer or by using the probe on the surface of the tooth.
  Score 2 = Moderate accumulation of soft deposits in the pocket, tooth or gingival margin, which can be seen without magnification.
  Score 3 = Abundance of soft material inside the bag and / or on the tooth and the gingival margin.
  The evaluation will be carried out in 4 points per tooth (disto-buccal, mesio-buccal, disto-palatal, mesio-palatal).
Chair time | During procedure
  The duration of the procedure will be timed, starting with the application of local anaesthesia and ending after the application of the bioactive material.
Patient satisfaction and perception | 1 week after baseline (regenerative intervention)
  - The presence or absence of bleeding, swelling, suppuration, tooth hypersensitivity and interference with daily activities will be assessed by dichotomous question. In case of a positive answer, 5-point Likert scale will be used (far too little, too little, about right, too much, far too much).
Patient satisfaction and perception | 1 week after baseline (regenerative intervention)
  Visual analog scale (VAS) will be used to evaluate the intensity of the discomfort and pain (Mounssif and cols., 2023). It consists of a horizontal line of 100 millimeters, with the extreme expressions of a symptom at each end. The left end represents absence or lower intensity, while the right end represents the highest intensity (Tonetti and cols., 2004). Patients are asked to mark on the line the point that indicates the intensity, and it is measured with a millimeter ruler. The intensity is expressed in millimeters. The assessment will be:
  * Mild pain if the patient scores pain as less than 30.
  * Moderate pain if the rating is between 40 and 70.
  * Severe pain if the rating is 80 or higher.
Patient satisfaction and perception | 1 week after baseline (regenerative intervention)
  - Oral health impact profile (OHIP-14, Spanish version). The OHIP-14 scores can range from 0 to 56 and are calculated by adding the ordinal values for each of the 14 domains. Scores for individual domains can range from 0 to 5 (Montero-Martín and cols., 2009).
Patient satisfaction and perception | 6 months after baseline (regenerative intervention)
  Patients will be asked to describe their perception of the outcome in terms of improvement in gingival bleeding, redness, gingival swelling, and hygiene capability. These parameters will also be measured using a Visual Analog Scale (VAS), where zero indicates no improvement and 100 indicates maximum improvement.
Patient satisfaction and perception | 12 months after baseline (regenerative intervention)
  Finally, the perception and satisfaction level with the aesthetic result of the treatment will be evaluated by selecting one of the following options: very satisfied, satisfied, neutral, moderately satisfied, or dissatisfied (Wismeyer and cols., 1995).

CONTACTS AND LOCATIONS:
Overall Officials: Andrés López Roldán, Study Director — University of Valencia; José Manuel Almerich Silla, Study Director — University of Valencia
Locations (1):
- Clínica Odontológica de la Universidad de Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Steffensen B, Webert HP. Relationship between the radiographic periodontal defect angle and healing after treatment. J Periodontol. 1989 May;60(5):248-54. doi: 10.1902/jop.1989.60.5.248. PMID 2738832
- [Background] Tonetti MS, Fourmousis I, Suvan J, Cortellini P, Bragger U, Lang NP; European Research Group on Periodontology (ERGOPERIO). Healing, post-operative morbidity and patient perception of outcomes following regenerative therapy of deep intrabony defects. J Clin Periodontol. 2004 Dec;31(12):1092-8. doi: 10.1111/j.1600-051X.2004.00615.x. PMID 15560811
- [Background] Anoixiadou S, Parashis A, Vouros I. Enamel matrix derivative as an adjunct to minimally invasive non-surgical treatment of intrabony defects: A randomized clinical trial. J Clin Periodontol. 2022 Feb;49(2):134-143. doi: 10.1111/jcpe.13567. Epub 2021 Nov 9. PMID 34708441
- [Background] Anoixiadou S, Parashis A, Vouros I. Minimally Invasive Non-Surgical Technique in the Treatment of Intrabony Defects-A Narrative Review. Dent J (Basel). 2023 Jan 11;11(1):25. doi: 10.3390/dj11010025. PMID 36661562